CLINICAL TRIAL: NCT02373852
Title: Post Marketing Surveillance (PMS) Retrospective Study of WIRION Performance in Patients Undergoing Saphenous Vein Graft (SVG) Intervention
Brief Title: PMS Retrospective Study of WIRION Performance in Patients Undergoing Saphenous Vein Graft (SVG) Intervention
Status: Completed | Type: Observational
Sponsor: Gardia Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SVG-CL003
Record Dates: First submitted 2014-09-22; First posted 2015-02-27 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Stenosis
MeSH Terms: conditions — Constriction, Pathologic | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Saphenous vein graft (SVG) stenting — Opening and stenting of blocked SVG with the use of the WIRION embolic protection filter

SUMMARY:
The objective of this study is to collect data on the use of the WIRION system in Patients undergoing Percutaneous Intervention of Saphenous Vein Graft (SVG).

DETAILED DESCRIPTION:
WIRION system is used as protection device in patients undergoing SVG stenting procedure. This retrospective study collects data on the usability of the WIRION during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent percutaneous intervention (PI) of SVG stenting in which the WIRIONTM system was used.
* Patient is greater than or equal to 18 years of age.

Exclusion Criteria:

* Undergone cardiac surgery in the past 60 days before the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing percutaneous intervention (PI) of saphenous vein graft (SVG) stenting
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vardit Segal, PhD, Study Director — Gardia medical manufacture the WIRION used in the study
Locations (1):
- Bnai Zion, Haifa, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- WIRION: Patients undergoing SVG stenting procedure with the use of the WIRION
Period: Overall Study
Arm/Group | WIRION
Started | 12 (Includes patients from a previous retrospective study NCT01042444)
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | WIRION
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 12
Diabetes [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events During the Procedure and up to 30 Days Following Procedure
Description: Collect and analyse all adverse events occurred during and following the SVG procedure up to 30 days.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | WIRION
Number analyzed (Participants) | 12
Participants | 5

2. Primary Outcome: Number of Patients That Undergo Successful SVG Procedure
Description: Successful procedure is considered as a procedure in which no distal embolization, dissection, perforation, abrupt closure or no reflow occurred.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | WIRION
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Arm/Group | WIRION
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WIRION (N=12)
Death (Cardiac disorders) | 1 — Cardiogenic shock
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WIRION (N=12)
Chest pain on effort (Cardiac disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No